CLINICAL TRIAL: NCT02257775
Title: Evolution of Resistance to Systemic Therapies in Patients With Breast Cancer
Acronym: EVOLUTION
Status: Terminated | Type: Observational
Why Stopped: Insufficient number of eligible and interested partients
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4203
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: n/a - observational

SUMMARY:
The objective of this study is to apply Whole-body DW imaging alongside the routine management of patients requiring systemic therapy for metastatic breast cancer to compare the time to progression of individual liver metastases within and between patients following stable disease or partial response to palliative systemic therapy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* First metastatic breast cancer relapse after treatment for early stage disease
* A minimum of 10 evaluable lesions in the liver on routine x-ray CT imaging
* Patient prescribed cytotoxic, endocrine or biological therapies
* Patient physically and psychologically fit enough to consider sequential WB-- - DWI imaging alongside their standard disease monitoring
* Written informed consent

Exclusion Criteria:

* Diagnosis of other cancer within the last 5 years, other than resected non-melanoma skin cancer or cervical intraepithelial neoplasia
* Diagnosis of brain metastases.
* Contraindication to magnetic resonance MR imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring systemic therapy for metastatic breast cancer
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Progression rate of liver metastases | 3 months
  Patients will be monitored by routine CT scans after 3 cycles of cytotoxic/biological therapy or after 3 months of endocrine therapy

SECONDARY OUTCOMES:
Progression rate of skeletal metastases | 3 months
  Patients will be monitored by routine CT scans after 3 cycles of cytotoxic/biological therapy or after 3 months of endocrine therapy
Global and local lesion Apparent Diffusion Coefficient (ADC) distributions of WB-DWI scans within individual patient | 3 months
  Patients will be monitored by routine CT scans after 3 cycles of cytotoxic/biological therapy or after 3 months of endocrine therapy
Patient acceptability of WB-DWI assessed from questionnaires provided between WB-DWI scans and quantified using a 5-point Likert scale | 3 months
  Patients will be monitored by routine CT scans after 3 cycles of cytotoxic/biological therapy or after 3 months of endocrine therapy
Comparison of patient acceptability to whole-body CT | 3 months
  Patients will be monitored by routine CT scans after 3 cycles of cytotoxic/biological therapy or after 3 months of endocrine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jill Noble, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden, Sutton, United Kingdom